CLINICAL TRIAL: NCT05823740
Title: Measuring Changes in Body Composition and Physical Function in Patients With Childhood Cancers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LCCC2232
Record Dates: First submitted 2023-04-10; First posted 2023-04-21 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Cancer; Malignant Neoplasm
Keywords: D3-creatine dilution method; pediatric; muscle mass; biological aging; physical function
MeSH Terms: conditions — Neoplasms | interventions — Hand Strength; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Other): Children with malignant diseases, receiving anti-cancer treatment and completed study interventions.
  Interventions: Other: Bioelectrical impedance Analysis (BIA); Other: D3-Creatine Dilution (D3Cr); Other: 6-Minute Walk Test (6MWT); Other: Timed Up and Go (TUG); Other: 30-second Sit-to-Stand (STS); Other: Hand Grip Strength (GS); Other: PBTL p16 expression; Other: CT, MR and PET Imaging

INTERVENTIONS:
Other: Bioelectrical impedance Analysis (BIA) — Bioelectrical impedance analysis (BIA) is a method for estimating body composition, in particular, body fat and muscle mass, where a weak electric current flows through the body and the voltage is measured in order to calculate the impedance (resistance) of the body. BIA will be done at baseline, during the study related to routine medical imaging, and end of the study.
Other: D3-Creatine Dilution (D3Cr) — The D3-Creatine dilution method is a safe and noninvasive measure of skeletal muscle mass that has previously been validated in adults, neonates, healthy children, and children. D3-Creatine Dilution will be done at baseline, during the study related to routine medical imaging, and end of the study.
Other: 6-Minute Walk Test (6MWT) — Cardiovascular fitness will be measured with the 6-minute walk test (6MWT). 6MWT will be done at baseline, during the study related to routine medical imaging, and end of the study.
Other: Timed Up and Go (TUG) — Balance and mobility will be assessed by the timed-up-and-go test (TUG). TUG will be done at baseline, during the study related to routine medical imaging, and end of the study.
Other: 30-second Sit-to-Stand (STS) — Strength and muscular function will be evaluated by modified 30-second sit-to-stand (STS). STS will be done at baseline, during the study related to routine medical imaging, and end of the study.
Other: Hand Grip Strength (GS) — Strength and muscular function will be evaluated by grip strength (GS). GS will be done at baseline, during the study related to routine medical imaging, and end of the study.
Other: PBTL p16 expression — Peripheral Blood biospecimen for PBTL p16 expression will be used for the assessment of biological aging. Blood biospecimens will be collected at baseline and end of the study for PBTL p16 analysis.
Other: CT, MR and PET Imaging — Participants will undergo routine imaging with either computed tomography (CT), Magnetic Resonance Imaging (MRI) of the chest or abdomen, or whole-body positron emission tomography (PET) scan. Skeletal muscle mass and fat mass will be calculated at several different vertebral levels from imaging studies.

SUMMARY:
The primary objective of this study is to evaluate the feasibility and acceptability of obtaining repeated measurements of lean muscle mass, physical function, and biological aging in children receiving active cancer therapy. The secondary objective is to evaluate the feasibility of using the D3-creatine dilution method (D3Cr) to measure skeletal muscle mass in children with cancer.

Assessments will be collected at diagnosis, once during active treatment, and end of treatment in coordination with routine imaging to monitor changes in study outcomes during active cancer treatment. Key sociodemographic, treatment and health-related factors will be abstracted from the medical record.

ELIGIBILITY:
Inclusion Criteria In order to participate in this study a subject must meet all of the eligibility criteria outlined below.

1. Ages 8-21 years at the time of cancer diagnosis
2. Must have a newly diagnosed malignant solid tumor or lymphoma.
3. Participant is expected to undergo cancer treatment with either chemotherapy, radiation, immunotherapy, or other biologically targeted therapy.
4. Participants will undergo routine imaging with either computed tomography (CT), or Magnetic Resonance Imaging (MRI) of the chest or abdomen, or whole-body positron emission tomography (PET) scan.
5. Written informed consent obtained to participate in the study and HIPAA authorization for the release of personal health information.
6. English or Spanish speaking
7. Subject is willing and able to comply with study procedures.
8. Since the patient is undergoing active cancer therapy, must obtain approval from the treating physician.

Exclusion Criteria All subjects meeting any exclusion criteria at baseline will be excluded from study participation.

1. Prior history of cancer
2. Treatment with surgical excision alone
3. Planned palliative treatment.
4. Subject has elected to forgo chemotherapy or radiotherapy.
5. Any diagnosis of leukemia.
6. Clinical concerns that the treating clinician feels would preclude participation in the study.
7. Subject has a pacemaker or bilateral joint prosthesis that would prevent undergoing BIA assessment.
8. Unwilling to sign informed consent.
9. Speak a language other than English or Spanish.

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
The feasibility of collecting body composition assessments | up to 12 months
  The feasibility of collecting body composition assessments will be measured as the % of participants completing all 3 assessments for each modality: D3-Creatine dilution method (D3Cr), Bioelectrical impedance Analysis (BIA), medical imaging (computerized tomography (CT), or magnetic resonance imaging (MRI), or positron emission tomography (PET).
The feasibility of collecting individual physical function assessments | up to 12 months
  The feasibility of collecting individual physical function assessments will be measured as the % of participants completing all 3 assessments for each modality namely the 6-Minute Walk Test (6MWT), Timed Up and Go (TUG), 30-second Sit-to-Stand (STS), Hand Grip Strength (GS)) at multiple time points during cancer therapy.

SECONDARY OUTCOMES:
Feasibility of collecting repeated measurements of biological aging (p16 expression) | up to 12 months
  The feasibility of collecting repeated measurements of biological aging (p16 expression) will be evaluated as % of participants completed both pre-treatment and post-treatment assessments.
The acceptability of the study | up to 12 months
  The acceptability of the study will be evaluated as the number of subjects approached and enrolled and number of subjects that withdraw from the study.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Smitherman, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data may be made available on an individual basis at the discretion of the PI.

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials